CLINICAL TRIAL: NCT01616134
Title: Effect of Korean Red Ginseng on Insulin Sensitivity in Non Diabetic Overweight Korean Adults
Acronym: KRGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Sang-Yeoup Lee, Pusan national iniversity Yangsan Hospital, The Korean Society of Ginseng
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: KRG-0912
Record Dates: First submitted 2012-06-05; First posted 2012-06-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Insulin Resistance; Obesity
Keywords: overweight,; ginseng
MeSH Terms: conditions — Insulin Resistance; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Korea Red Ginseng (Active Comparator): Intervention group were administered with 4 capsules (2 g) each of powdered red ginseng (6-year old , rootlets) 40 minutes before breakfast, lunch and dinner, totaling 12 capsules (6 g) per day, for 12 weeks.
  Interventions: Other: Korea red ginseng
- placebo contating constarch (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Korea red ginseng — Intervention group were administered with 4 capsules (2 g) each of powdered red ginseng (6-year old , rootlets) 40 minutes before breakfast, lunch and dinner, totaling 12 capsules (6 g) per day, for 12 weeks
  Arms: Korea Red Ginseng
Other: Placebo — The subjects in the Control group were given the same quantity of placebos also three times a day for 12 weeks.
  Arms: placebo contating constarch

SUMMARY:
Korean red ginseng (KRG) is popular worldwide since it is believed to contain ingredients with a variety of health enhancement effects. Several in vitro studies and animal studies showed that ginseng has anti-obesity, anti-diabetic and anti-metabolic disease effects. Several studies involving type 2 diabetes mellitus (T2DM) patients reported that administration of KRG for 12 weeks resulted in positive effects on the maintenance of sugar control effect and improvement of insulin resistance Although there is evidence to suggest that KRG could efficacious reduction in postprandial glycemia, the benefits of long-term KRG in healthy individuals on insulin sensitivity has not yet been established. Therefore, we investigated whether KRG affected insulin sensitivity in healthy overweight or obese Korean subjects without overt diabetes.

DETAILED DESCRIPTION:
80 adults between the ages of 20 and 60 years and with a BMI ≥ 23 kg/m2 was initially enrolled. The subjects had not taken any supplements or medications, including anti-diabetic drugs, anti-hypertensive drugs, steroids, or hormonal products, during the previous 4 weeks.

This study had a randomized, placebo-controlled, double-blind controlled design. Each subject was randomized to either the Intervention group or the Control group. The subjects in the Intervention group were administered with 4 capsules (2 g) each of powdered red ginseng (6-year old , rootlets) 40 minutes before breakfast, lunch and dinner, totaling 12 capsules (6 g) per day, for 12 weeks. The subjects in the Control group were given the same quantity of placebos also three times a day for 12 weeks.

Blood samples after a 12-h fast were taken at baseline and 12 weeks after randomization. Blood samples were taken after at least 8 hours of fasting for general blood test, biochemical test and lipid test. Each subject's diet was monitored by a semi-quantitative FFQ at baseline and after 12 weeks. Participants were asked to report the frequency of consumption of 53 food items contained in the semi-quantitative FFQ over the 2 weeks prior to administration by an experienced dietitian. Excessive drinking was defined according to the guidelines of the National Institute Alcohol Abuse and Alcoholism when more than 14 glasses (alcohol 196 g) are consumed for male and 7 glasses (alcohol 98 g) for female. Physical activity was assessed using the International Physical Activity Questionnaire at baseline and after 12 weeks. We expressed physical activity levels as MET-minute. METs are multiples of the resting metabolic rates. A MET-minute is computed by multiplying the MET score of an activity by the minutes performed. MET-minute scores are equivalent to kilocalories for a 60 kilogram person.

ELIGIBILITY:
Inclusion Criteria:

* ages of 20 and 60 years
* BMI ≥ 23 kg/m2

Exclusion Criteria:

* any supplements or medications, including anti-diabetic drugs, anti-hypertensive drugs, steroids, or hormonal products, during the previous 4 weeks
* participant's systolic BP was above 140 mmHg or diastolic BP above 90 mmHg
* above 100 m/dL before enrollment in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity (insulin, HOMA-IR, QUICKI) | 12 weeks
  Blood samples after a 12-h fast were taken at baseline and 12 weeks after randomization. Blood samples were taken after at least 8 hours of fasting for glucose, insulin, liver enzyme, creatinine and lipid test. The homeostasis model assessment index-insulin resistance (HOMA-IR) was calculated using a fomula: [fasting plasma insulin (µU/mL) × fasting plasma glucose (mg/dL)] / (22.5×18.182) and quantitative insulin-sensitivity check index (QUICKI) was calculated using a formula: 1 / [log fasting insulin (µU/mL) + log fasting blood sugar (mg/dL)]

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea